CLINICAL TRIAL: NCT03539692
Title: Prescreening Protocol to Enroll in Food Allergy Clinical Studies at a Single Site
Acronym: Prescreen
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Sayantani B. Sindher, Clinical Assistant Professor, Stanford University
Other Study IDs: 34738; 1UM1AI130839-01 (NIH); FY20ITN384 (Other Grant/Funding Number: NIH Prime Immune Tolerance Network); 5U19AI104209-07 (NIH); 5UM1AI82034-02 (Other Grant/Funding Number: NIH Prime Johns Hopkins University)
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-05

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood will be collected, additional samples could include sputum, saliva, urine sample, stool sample, oral and nasal samples, skin samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a protocol for prescreening of participants who would like to be in clinical studies in our Center at Stanford.

ELIGIBILITY:
Inclusion Criteria:

* Any individual with possible food allergy (as per their clinical history) who is interested in performing the gold standard food challenge for diagnosis.

Exclusion Criteria:

* Any individual who does not consent
* Any individual who is currently taking oral steroids
* Any individual with moderate to severe asthma (FEV1<80%)

Ages: 1 Week to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ages 1 wk-90 yrs will be screened and enrolled in this study to determine if they have a clinically-relevant food allergy. If so, they could be eligible for interventional clinical trials in the future.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-06-10 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Outcome of standardized food challenges | 1 year
  Standardized Oral food challenges will occur in a staged manner to diagnose food allergies

SECONDARY OUTCOMES:
skin testing will occur to evaluate food allergen responses | 1 year
  Standardized skin testing will be performed to detect sensitivity to food allergens

CONTACTS AND LOCATIONS:
Overall Officials: Sayantani Sindher, MD, Principal Investigator — Stanford University, SNP Center for Food Allergy and Asthma Research
Locations (1):
- The Sean N. Parker Center for Allergy and Asthma Research, Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Purington N, Chinthrajah RS, Long A, Sindher S, Andorf S, O'Laughlin K, Woch MA, Scheiber A, Assa'ad A, Pongracic J, Spergel JM, Tam J, Tilles S, Wang J, Galli SJ, Desai M, Nadeau KC. Eliciting Dose and Safety Outcomes From a Large Dataset of Standardized Multiple Food Challenges. Front Immunol. 2018 Sep 21;9:2057. doi: 10.3389/fimmu.2018.02057. eCollection 2018. PMID 30298065